CLINICAL TRIAL: NCT06182358
Title: Randomized Controlled Trial to Evaluate the Impact of XDEMVY® on Demodex Blepharitis in Soft Contact Lens Wearers
Brief Title: Impact of XDEMVY® on Demodex Blepharitis in Soft Contact Lens Wearers
Acronym: Ariel
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Tarsus Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: TRS-023
Record Dates: First submitted 2023-12-13; First posted 2023-12-26 (Actual); Last update posted 2025-07-02 (Actual); Status verified 2025-06

CONDITIONS: Demodex Blepharitis
Keywords: Soft contact lenses

STUDY DESIGN:
Intervention Model Description: Active arm: XDEMVY 0.25% Control arm: Vehicle of XDEMVY
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Treatment assignment will be unknown to the study participants, investigators, and site staff performing study assessments
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- Active Treatment (Experimental): XDEMVY (lotilaner ophthalmic solution) 0.25%, administered topically twice a day for approximately 43 days
  Interventions: Drug: Lotilaner ophthalmic solution, 0.25%
- Control (Placebo Comparator): Vehicle of XDEMVY ophthalmic solution, administered topically twice a day for approximately 43 days
  Interventions: Drug: Vehicle control

INTERVENTIONS:
Drug: Lotilaner ophthalmic solution, 0.25% — XDEMVY (lotilaner ophthalmic solution) 0.25%, administered topically twice a day for approximately 43 days
  Arms: Active Treatment
Drug: Vehicle control — Vehicle of XDEMVY administered topically twice a day for approximately 43 days
  Arms: Control

SUMMARY:
To compare the efficacy of XDEMVY ophthalmic drop to its vehicle control for the treatment of Demodex blepharitis and its impact on the soft contact lens wearing experience.

DETAILED DESCRIPTION:
This Phase 4 study is a prospective, multicenter, randomized, vehicle-controlled, double-masked, two-arm, parallel treatment clinical trial of participants who have Demodex blepharitis and are current daily wear soft contact lenses wearers. The primary outcome measure is the reduction of collarettes at Day 43. The secondary outcome measures are the reduction of eyelid margin erythema at Day 43; subject-reported comfortable contact lens daily wear time; and total contact lens wear time. Safety will be determined by assessing adverse effects related to study drug administration as well as evaluating any clinically significant changes from baseline in visual acuity and slit lamp biomicroscopy findings.

ELIGIBILITY:
Inclusion Criteria:

* Be willing to sign the informed consent form and is deemed capable of complying with the requirements of the study protocol
* Must meet the following criteria in at least one eye: Have more than 10 eyelashes (Grade 2 or higher) with collarettes on the upper or lower eyelid; have at least Grade 1 erythema of the lower eyelid; and have a total meibomian gland secretion score ≥ 12 but ≤ 32 AND have a minimum of 6 expressible glands for the 15 glands evaluated on the lower eyelid
* Currently wearing soft contact lenses on both eyes an average of at least 2 days per week with an average minimum wearing time of 6 hours each day over the past 3 months and is able and willing to continue to wear contact lenses during the study

Exclusion Criteria:

* Use of artificial tears or rewetting drops within 24 hours of the Screening visit or unwilling to forego the use of this treatment during the study
* Prescription AND systemic, drug delivery implant, ocular topical, or topical: antibacterial, anti-parasitic, or anti-inflammatory corticosteroid treatment within 14 days of the Screening or Day 1 visits
* Use of TYRVAYA™ Nasal Spray (varenicline solution, Oyster Point Pharma) within 14 days of the Screening visit or unwilling to forego the use of this treatment during the study
* Use of XDEMVY™ (lotilaner ophthalmic solution) 0.25%, Tarsus Pharmaceuticals, Inc., within 12 months of the Screening visit
* Treatment for blepharitis (e.g., tea tree oil-based products, hypochlorous acid-based products, commercial eyelid foams, eyelid wipes, lid scrubs, etc.) within 14 days of the Screening visit or unwilling to forego the use of these treatments during the study
* Use of artificial eyelashes or eyelash extensions at the Screening visit if they limit accurate eyelid margin assessment
* Currently pregnant or lactating

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 145 (Actual)
Dates: Start 2023-12-27 (Actual); Primary Completion 2025-01-27 (Actual); Study Completion 2025-01-27 (Actual)

PRIMARY OUTCOMES:
Reduction of collarettes at Day 43 | 43 days
  Change in collarette score at Day 43 compared to baseline, graded from 0 (0 to 2 lashes have collarettes per eyelid) to 4 ( 2/3 or more of lashes have collarettes per eyelid)

SECONDARY OUTCOMES:
Reduction of eyelid margin erythema at Day 43 | 43 days
  Change in eyelid margin erythema score at Day 43 compared to baseline, graded from 0 (normal) to 3 (severe)
Subject-reported comfortable daily wear time | 43 days
  Comfortable daily wear time in hours per day
Total contact lens wear time | 43 days
  Total daily wear time in hours per day

CONTACTS AND LOCATIONS:
Overall Officials: Blake Simmons, OD, Principal Investigator — Vision Institute
Locations (14):
- United States (14):
  - Site, Cave Creek, Arizona
  - Site, Long Beach, California
  - Vision Institute, Colorado Springs, Colorado
  - Site, Delray Beach, Florida
  - Site, Indianapolis, Indiana
  - Site, Pittsburg, Kansas
  - Site, Louisville, Kentucky
  - Site, Edina, Minnesota
  - Site, Shelby, North Carolina
  - Site, Fargo, North Dakota
  - Site, Powell, Ohio
  - Site, Cranberry Township, Pennsylvania
  - Site, Memphis, Tennessee
  - Site, Houston, Texas

IPD SHARING:
Plan to Share IPD: No